CLINICAL TRIAL: NCT04596475
Title: Prevention of Transmission of Hepatitis C Virus (HCV) From HCV-Viremic Organ Donor to HCVNegative Organ Transplant Recipient - Pilot Trial
Brief Title: Prevention of Transmission of Hepatitis C Virus (HCV) From HCV-Viremic Organ Donor
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Saima Aslam, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Project #200895
Record Dates: First submitted 2020-09-28; First posted 2020-10-22 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis C; Hepatitis C Virus Infection, Response to Therapy of
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir; pibrentasvir

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: glecaprevir/pibrentasvir (GLE/PIB)

INTERVENTIONS:
Drug: glecaprevir/pibrentasvir (GLE/PIB) — The study intervention consists of a single daily dose of GLE/PIB 100/40 mg (one dose consists of 3 tablets) administered orally; or crushed and administered via a feeding tube if participant is unable to swallow by mouth, for example in the immediate post-operative period. First dose will be administered in the pre-operative period within 4 hours of surgery followed by once daily doses for 7 days total.

SUMMARY:
This trial will be done in participants who undergo transplantation of heart, kidney or lung at University of California, San Diego (UCSD) and receive a hepatitis C infected donor organ. In this trial, the plan is to start hepatitis C treatment just before transplant surgery and treat for a short one-week course to see if hepatitis C infection can be prevented in the transplant recipient. The plan is to perform this trial in 10 participants and if successful, the next step is to try to make it standard of care as prevention of infection is better than treating hepatitis C after discharge from transplant surgery (which is usually a 12 week standard treatment).

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years or greater
* participants actively listed for heart, lung and/or kidney transplant
* participants have already consented to receive HCV-viremic organs as part of the institution's clinical practice protocol (involves education and informed consent), and are able to sign informed consent for this research study.

Exclusion Criteria:

* participants who have a prior history of HCV infection regardless of treatment status, pre-existing human immunodeficiency virus (HIV) or hepatitis B virus (HBV) infection
* participants who are not able to sign informed consent for this research study
* participants who have not agreed to accept HCV+ organs as part of the UCSD clinical practice protocol
* participants who are listed for a liver transplant (either as a single organ or combined organ transplant).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with Sustained Virological Response | 91 days
  The primary outcome is the percentage of patients sustained virological response (SVR) at day 91 after completion of a 7-day course of GLE/PIB.

SECONDARY OUTCOMES:
Percentage of participants with treatment-related Serious Adverse Events | 91 days
  Safety and tolerability of the 7-day GLR/PIB course. Safety and tolerability will be assessed by documenting Serious Adverse Events (based on NIH criteria) for the duration of the study. Safety assessments will occur through review of the medical record of the patient, review of laboratory parameters and open-ended questions at the in-person assessments.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, San Diego, California, United States

REFERENCES:
- [Background] Aslam S, Yumul I, Mariski M, Pretorius V, Adler E. Outcomes of heart transplantation from hepatitis C virus-positive donors. J Heart Lung Transplant. 2019 Dec;38(12):1259-1267. doi: 10.1016/j.healun.2019.08.019. Epub 2019 Aug 24. PMID 31521479
- [Background] Bethea ED, Gaj K, Gustafson JL, Axtell A, Lebeis T, Schoenike M, Turvey K, Coglianese E, Thomas S, Newton-Cheh C, Ibrahim N, Carlson W, Ho JE, Shah R, Nayor M, Gift T, Shao S, Dugal A, Markmann J, Elias N, Yeh H, Andersson K, Pratt D, Bhan I, Safa K, Fishman J, Kotton C, Myoung P, Villavicencio MA, D'Alessandro D, Chung RT, Lewis GD. Pre-emptive pangenotypic direct acting antiviral therapy in donor HCV-positive to recipient HCV-negative heart transplantation: an open-label study. Lancet Gastroenterol Hepatol. 2019 Oct;4(10):771-780. doi: 10.1016/S2468-1253(19)30240-7. Epub 2019 Jul 26. PMID 31353243
- [Background] Kwong AJ, Wall A, Melcher M, Wang U, Ahmed A, Subramanian A, Kwo PY. Liver transplantation for hepatitis C virus (HCV) non-viremic recipients with HCV viremic donors. Am J Transplant. 2019 May;19(5):1380-1387. doi: 10.1111/ajt.15162. Epub 2018 Nov 26. PMID 30378723
- [Background] Woolley AE, Singh SK, Goldberg HJ, Mallidi HR, Givertz MM, Mehra MR, Coppolino A, Kusztos AE, Johnson ME, Chen K, Haddad EA, Fanikos J, Harrington DP, Camp PC, Baden LR; DONATE HCV Trial Team. Heart and Lung Transplants from HCV-Infected Donors to Uninfected Recipients. N Engl J Med. 2019 Apr 25;380(17):1606-1617. doi: 10.1056/NEJMoa1812406. Epub 2019 Apr 3. PMID 30946553
- [Background] Gupta G, Yakubu I, Bhati CS, Zhang Y, Kang L, Patterson JA, Andrews-Joseph A, Alam A, Ferreira-Gonzalez A, Kumar D, Moinuddin IK, Kamal L, King AL, Levy M, Sharma A, Cotterell A, Reichman TW, Khan A, Kimball P, Stiltner R, Baldecchi M, Brigle N, Gehr T, Sterling RK. Ultra-short duration direct acting antiviral prophylaxis to prevent virus transmission from hepatitis C viremic donors to hepatitis C negative kidney transplant recipients. Am J Transplant. 2020 Mar;20(3):739-751. doi: 10.1111/ajt.15664. Epub 2019 Nov 15. PMID 31652392
- [Background] Aslam S, Grossi P, Schlendorf KH, Holm AM, Woolley AE, Blumberg E, Mehra MR; working group members. Utilization of hepatitis C virus-infected organ donors in cardiothoracic transplantation: An ISHLT expert consensus statement. J Heart Lung Transplant. 2020 May;39(5):418-432. doi: 10.1016/j.healun.2020.03.004. Epub 2020 Mar 19. PMID 32362393